CLINICAL TRIAL: NCT04170712
Title: Data and Specimen Bank of Patients Diagnosed With, and at High-risk for, Gynecologic Cancers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Sponsor
Other Study IDs: 18620
Record Dates: First submitted 2019-11-17; First posted 2019-11-20 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Ovarian Cancer
Keywords: tampons; ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tampons, swabs, blood and tissue will be collected prospectively to establish a bank of samples fro future testing for markers, risk factors and targets for ovarian cancer prevention, detection and treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgical or High Risk: Patients with confirmed diagnosis of ovarian cancer or suspicious mass or who have a family history or genetic mutation that puts them at high risk fro ovarian cancer.
  Interventions: Other: Tampons

INTERVENTIONS:
Other: Tampons — Collection of tampons, blood, cervical swabs, tissue and ascites

SUMMARY:
The purpose of this project is to establish a bank at UVa of tampon samples, cervical swabs, blood, associated tumor specimens that would otherwise be discarded, and relevant medical data from consenting patients that have suspected and/or confirmed gynecological cancer diagnoses. The specimens collected will be saved for analysis on future projects to determine if factors in the specimens are predictive and/or correlated to gynecological cancer diagnoses and/or outcomes

DETAILED DESCRIPTION:
The purpose of this project is to establish a bank at UVa of tampon samples, cervical swabs, blood, associated tumor specimens that would otherwise be discarded, and relevant medical data from consenting patients that have suspected and/or confirmed gynecological cancer diagnoses. The specimens collected will be saved for analysis on future projects to determine if factors in the specimens are predictive and/or correlated to gynecological cancer diagnoses and/or outcomes. The bank will contain: 1) 10cc of blood drawn through venipuncture annually; 2) tampons placed in the patients vagina prior to surgery or clinic visit; 3) swabs of the endocervical canal; 4) freshly collected leftover and to-be-discarded tumors from ovarian, uterine, cervical, as well as leftover normal tissue, and ascites fluid, from samples collected for diagnostic purposes. These samples and patient-associated medical record data will be banked and used for future research and analyses. Samples will be saved in multiple formats for later tumor profiling (i.e. FFPE, snap frozen, in RNA-later, etc). These samples and information will be used to determine the underlying causes of cancers and chemoresistance, so that better methods of treatment, management, and prevention of gynecological cancers may be discovered in the future.

Samples will be linked and coded, with all HIPAA protected information removed, for storage and sharing with other investigators to protect patient information. Only coded samples and clinical information will be used in this protocol for when samples, information, and/or data are shared with other investigators at UVa or outside institutions in the future. A separate password protected/encrypted file will contain the patient identifiers and the key to the coded sample numbers. This file will only be accessible by the PI or study team listed on this protocol on UVa premises, and will only be stored on a UVa server behind the UVa firewall, and will not be stored or accessed on personal computers. Thus, identified patient information will not be accessible to any individual, except the PI or study team listed on this protocol, ensuring protection of patient information. In addition, coded patient samples and medical data from specimens obtained from the University of Alabama-Birmingham, that were previously collected by the PI under local IRB approval (IRB-HSR #18042), have been transferred to UVA under a fully executed MTA, and will be assimilated into this databank at UVa for future research.

ELIGIBILITY:
Inclusion Criteria:

* Adult female non-pregnant patients with high risk for gynecological and/or breast cancer who will be:

  * undergoing a planned surgery with the UVa Department of gynecological oncology for gynecological, breast, and/or related cancers and conditions
  * undergoing surveillance in the high-risk gynecological oncology clinic for gynecological, breast, and/or related cancers and conditions

Exclusion Criteria:

* • Is under the age of 18

  * is pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients with confirmed ovarian cancer diagnosis or suspicious mass or patients with a strong family history of ovarian cancer or genetic mutation that puts them at high risk for ovarian cancer
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2016-06-10 (Actual); Primary Completion 2022-06-10 (Estimated); Study Completion 2022-06-10 (Estimated)

PRIMARY OUTCOMES:
To establish a bank of specimens at UVa | 10 years
  banking specimens for future testing

CONTACTS AND LOCATIONS:
Overall Officials: Charles Landen, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No